CLINICAL TRIAL: NCT00174239
Title: A Double-Blind, Randomized, Comparative Study of Cabaser and Sinemet CR For The Treatment Of Nocturnal Disability In Levodopa -Treated Parkinson's Disease Patients.
Brief Title: Study Of Cabaser and Sinemet CR For The Treatment Of Nighttime Symptoms Associated With Parkinson's Disease.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A7231001
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Cabergoline; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cabergoline
Drug: controlled-release levodopa / carbidopa

SUMMARY:
The study will assess the relative benefit of cabergoline vs carbidopa/levodopa therapy in treating nighttime problems of Parkinson Disease.

DETAILED DESCRIPTION:
The trial was terminated prematurely June 26, 2005 due to the inability to re-supply study drug for the planned number of subjects. There were no safety or efficacy concerns regarding the study in the decision to terminate the trial.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson Disease
* Must be experiencing sleep akinesia

Exclusion Criteria:

* Current treatment with other dopamine agonists
* Nocturnal hallucinations
* Dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-07; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
PDSS, UPDRS

SECONDARY OUTCOMES:
CGI, PGI, Epworth Sleepiness Scale, PDQ-39

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Australia (2):
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Brisbane, Queensland
- Italy (8):
  - Pfizer Investigational Site, Loc. Camerelle - Pozzilli, IS
  - Pfizer Investigational Site, Vittoria, Ragusa
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Bolzano
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Padua
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Roma
- Spain (4):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7231001&StudyName=Study+Of+Cabaser+and+Sinemet+CR+For+The+Treatment+Of+Nighttime+Symptoms+Associated+With+Parkinson%27s+Disease%2E